CLINICAL TRIAL: NCT05365984
Title: Study on the Intelligent Follow-up Management Model of Neonatal Jaundice After Discharge Based on Early Multi-dimensional Indicators and Internet Communications
Brief Title: Intelligent Follow-up of Neonatal Jaundice Based on Early Indicators and Internet Communications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); Jiaxing University Affiliated Women and Children Hospital (Unknown); Ningbo Women & Children's Hospital (Other); Shaoxing Women's and Children's Hospital (Unknown); Jinhua Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRO2021-1366
Record Dates: First submitted 2022-04-15; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-04

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: End tidal carbon monoxide; Internet Plus; jaundice follow-up management model
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal | interventions — Technology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- innavative modeled strategy (Experimental): In this arm, the risk evaluation before discharge for hyperbilirubenemia needing further intervention is based on Bhutani nomogram and end tidal carbon monoxide corrected for ambient carbon monoxide. Assessment result includes high risk, median risk, low risk and delayed discharge. Internet Plus technology is applied in follow-up management.
  Interventions: Diagnostic Test: end tidal carbon monoxide corrected for ambient carbon monoxide （ETCOc）; Other: Internet Plus technology
- traditional strategy (No Intervention): In this arm, the risk evaluation before discharge for hyperbilirubenemia needing further intervention is based on Bhutani nomogram and the follow-up table advised by the Chinese guideline for neonatal hyperbilirubinemia. Assessment result includes high risk, median risk and low risk. Traditional outpatient is applied in follow-up management.

INTERVENTIONS:
Diagnostic Test: end tidal carbon monoxide corrected for ambient carbon monoxide （ETCOc） — The measurement of end tidal carbon monoxide corrected for ambient carbon monoxide （ETCOc）is conducted in the process of risk evaluation.
  Arms: innavative modeled strategy
Other: Internet Plus technology — The Internet Plus technology is applied in the process of follow-up management.
  Arms: innavative modeled strategy

SUMMARY:
In this prospective multi-center randomized clinical trial, a new follow-up strategy for neonatal jaundice after discharge will be evaluated. It is based on current risk factors of neonatal hyperbilirubinemia, added with the rate of bilirubin production (exhaled carbon monoxide measurement) as a new indicator,and incorporated with Internet Plus technology. Traditional methods following the Chinese guideline for neonatal hyperbilirubinemia were applied in the control group. The morbidity of BIND, the number of outpatient follow-up after discharge and the convenience will be compared between the two groups. The accuracy, effectiveness, safety and convenience of the study strategy will be testified.

DETAILED DESCRIPTION:
The eligible newborns will be randomized into two groups: the study group (innovative strategy) and the controlled group (traditional strategy).

The innovative strategy included the ETCOc measurement in the risk evaluating process and the Internet Plus approach in the follow-up process.

ELIGIBILITY:
Inclusion Criteria:

1. gestational age between 35(+0)~41(+6)
2. birth weight ≥ 2500 g
3. ethics approval obtained
4. parental consent obtained

Exclusion Criteria:

1. severe perinatal asphyxia
2. infectious diseases
3. persistent need for respiratory support
4. major congenital malformation
5. inborn errors of metabolism
6. pathological neonatal hyperbilirubinemia due to the defects of red blood cell membrane and erythrocyte enzyme

Ages: 12 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2500 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of acute bilirubin encephalitis | within 2 week after birth
  the number of infants with acute bilirubin encephalitis in each group
the bilirubin level of readministration for hyperbilirubinemia | within 1 months
  the average bilirubin level of infants, who are readmitted for hyperbilirubinemia

SECONDARY OUTCOMES:
the cost for the issue of jaundice follow-up | within 1 month
  compare the fee for intelligent follow-up with the fee for clinical visiting according to present jaundice follow-up suggestion
the time for the issue of jaundice follow-up | within 1 month
  compare the time for intelligent follow-up，including the time for TSB measurement and internet commuication，with the time for clinical visiting according to present jaundice follow-up suggestion

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhu, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhutani VK, Wong RJ, Stevenson DK. Hyperbilirubinemia in Preterm Neonates. Clin Perinatol. 2016 Jun;43(2):215-32. doi: 10.1016/j.clp.2016.01.001. Epub 2016 Mar 23. PMID 27235203
- [Background] Cortey A, Renesme L, Raignoux J, Bedu A, Casper C, Tourneux P, Truffert P. [Management of jaundice in the newborn>/=35 GW: From screening to follow-up after discharge. Guidelines for clinical practice]. Arch Pediatr. 2017 Feb;24(2):192-203. doi: 10.1016/j.arcped.2016.11.011. Epub 2017 Jan 14. French. PMID 28094087
- [Background] Du L. [Prevention and intervention strategies for hyperbilirubinemia induced brain injury]. Zhonghua Er Ke Za Zhi. 2014 Oct;52(10):721-3. No abstract available. Chinese. PMID 25537534
- [Background] Castillo A, Grogan TR, Wegrzyn GH, Ly KV, Walker VP, Calkins KL. Umbilical cord blood bilirubins, gestational age, and maternal race predict neonatal hyperbilirubinemia. PLoS One. 2018 Jun 1;13(6):e0197888. doi: 10.1371/journal.pone.0197888. eCollection 2018. PMID 29856776
- [Background] Bhutani VK, Maisels MJ, Schutzman DL, Castillo Cuadrado ME, Aby JL, Bogen DL, Christensen RD, Watchko JF, Wong RJ, Stevenson DK. Identification of risk for neonatal haemolysis. Acta Paediatr. 2018 Aug;107(8):1350-1356. doi: 10.1111/apa.14316. Epub 2018 Apr 16. PMID 29532503
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Background] Subspecialty Group of Neonatology, The Society of Pediatrics, Chinese Medical Association. [The experts consensus on the management of neonatal hyperbilirubinemia]. Zhonghua Er Ke Za Zhi. 2014 Oct;52(10):745-8. No abstract available. Chinese. PMID 25537539
- [Background] Rong ZH, Luo F, Ma LY, Chen L, Wu L, Liu W, Du LZ, Luo XP. [Evaluation of an automatic image-based screening technique for neonatal hyperbilirubinemia]. Zhonghua Er Ke Za Zhi. 2016 Aug;54(8):597-600. doi: 10.3760/cma.j.issn.0578-1310.2016.08.008. Chinese. PMID 27510872
- [Background] Tabatabaee RS, Golmohammadi H, Ahmadi SH. Easy Diagnosis of Jaundice: A Smartphone-Based Nanosensor Bioplatform Using Photoluminescent Bacterial Nanopaper for Point-of-Care Diagnosis of Hyperbilirubinemia. ACS Sens. 2019 Apr 26;4(4):1063-1071. doi: 10.1021/acssensors.9b00275. Epub 2019 Mar 29. PMID 30896150
- [Background] Dalal SS, Mishra S, Agarwal R, Deorari AK, Paul V. Does measuring the changes in TcB value offer better prediction of Hyperbilirubinemia in healthy neonates? Pediatrics. 2009 Nov;124(5):e851-7. doi: 10.1542/peds.2008-3623. Epub 2009 Oct 12. PMID 19822593
- [Background] Ma X, Zhu J, Du L. Neonatal Management During the Coronavirus Disease (COVID-19) Outbreak: The Chinese Experience. Neoreviews. 2020 May;21(5):e293-e297. doi: 10.1542/neo.21-5-e293. No abstract available. PMID 32358142
- [Background] Ma XL, Chen Z, Zhu JJ, Shen XX, Wu MY, Shi LP, Du LZ, Fu JF, Shu Q. Management strategies of neonatal jaundice during the coronavirus disease 2019 outbreak. World J Pediatr. 2020 Jun;16(3):247-250. doi: 10.1007/s12519-020-00347-3. Epub 2020 Feb 28. PMID 32112336